CLINICAL TRIAL: NCT03372837
Title: A Multicenter, Open-label Phase III Study of SyB L-0501 in Combination With Rituximab in Patients With Recurrent or Relapsed Diffuse Large B-Cell Lymphoma
Brief Title: Phase III Study of SyB L-0501 in Combination With Rituximab to Treat Recurrent/Relapsed Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017002
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-06

CONDITIONS: Assess the Efficacy and Safety of SyB L-0501 in Combination With Rituximab in Patients With Recurrent or Relapsed DLBCL
Keywords: Diffuse large B-cell lymphoma, rituximab, SyB L-0501, combination therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SyB L-0501 (Experimental): The administration of SyB L-0501 at 120 mg/m^2/day by intravenous infusion on Day 2 and Day 3 of each 21-day cycle with up to 6 cycles. Dose modifications are permitted from 2nd cycle according to dose reduction schedule.
  SyB L-0501 60 mg/m^2, 90 mg/m^2 or 120 mg/m^2/day on Day 2 and Day 3 will be followed by 18 days of observation.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — The administration of rituximab at 375 mg/m^2/day by intravenous infusion on Day 1 of each 21-day cycle with up to 6 cycles. Dose modifications are not permitted.

SUMMARY:
The purpose of this study is to determine the efficacy of SyB L-0501 in combination with rituximab in patients with recurrent/relapsed diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Primary Objective is to determine the efficacy, as measured by overall response rate on the basis of Revised Response Criteria for Malignant Lymphoma, of SyB L-0501 at 120 mg/m^2/day on Day 2 and Day 3 in combination with rituximab at 375 mg/m^2 on Day 1 of each 21-day cycle in patients with recurrent/relapsed diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion criteria Patients who satisfy all of the conditions listed below.

1. Patients with histopathologically confirmed diffuse large B-cell lymphoma (DLBCL) except for transformed lymphoma on the basis of World Health Organization (WHO) histological classification (4th ed., 2008).
2. Patients with documented Cluster of differentiation 20 (CD20)-positive for lymphoma cells.
3. Patient with recurrent or relapsed DLBCL after R-CHOP-like theraphy as the firstline therapy.
4. Patients with measurable lesions >1.5 cm in major axes.
5. Patients who are expected to survive for at least 3 months.
6. Patients aged 20 or above at the time informed consent is obtained.
7. Patient with Performance Status (P.S.) 0-1.
8. Patients with adequately maintained organ function.

Exclusion Criteria The study subject should be excluded if any one of the following condition exists.

1. Patients who have been without treatment for less than 3 weeks after prior treatment.
2. Patients who can be candidates for autologous peripheral blood stem cell transplantation at the discretion of the investigator.
3. Patients who received adequate prior treatments and did not respond to any of them.
4. Patient who received prior chemotherapy 3 regimens or more.
5. Patients with central nervous system (CNS) involvement or patients with clinical symptoms suggestive of CNS involvement.
6. Patient with serious active infection.
7. Patient with serious complication.
8. Patient with complication or medical history of serious cardiac disease.
9. Patient with serious gastrointestinal symptoms.
10. Patient with malignant pleural effusion, pericardial effusion, or ascites retention.
11. Patients positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or HIV antibody.
12. Patient with serious bleeding tendency.
13. Patient with a fever of 38.0°C or higher.
14. Patients with, or confirmed in the past to have had, interstitial pneumonia, pulmonary fibrosis, or pulmonary emphysema.
15. Patients with active multiple primary cancer or patients with a history of other malignant cancer within the past 5 years, except for basal cell cancer of the skin, squamous cell cancer, or cervical cancer in situ.
16. Patients with, or confirmed in the past to have had, autoimmune hemolytic anemia.
17. Patient who received bendamustin hydrochloride in the past.
18. Patients who received cytokine preparation such as erythropoietin or granulocyte colony-stimulating factor (G-CSF) or blood transfusions within 2 weeks before the examination at registration for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | up to 30 weeks
  Complete Response (CR) + Partial Response (PR) Determined on the Basis of Revised Response Criteria for Malignant Lymphoma (Revised RC 2007)

SECONDARY OUTCOMES:
Complete Response (CR) Rate | up to 30 weeks
  Determined on the Basis of Revised Response Criteria for Malignant Lymphoma (Revised RC 2007)
Progression Free Survival (PFS) | up to 30 weeks
  PFS = day of the first PFS event - day of start of study treatment + 1
Duration of Response (DOR) | up to 30 weeks
  DOR is the period from the date of achieving CR, or PR in the responders to the earliest onset date of any progression events calculated using the Kaplan-Meier estimator. The median and the 95% Confidence Interval (CI ) were calculated using Greenwood's formula.
Overall Survival (OS) | up to 30 weeks.
  Death due to any given cause was defined as an event. OS was calculated using the Kaplan-Meier estimator. The median and the 95% CI were calculated using Greenwood's formula.

CONTACTS AND LOCATIONS:
Locations (29):
- Japan (29):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyoake, Aichi-ken
  - Research Site, Matsuyama, Ehime
  - Research Site, Maebashi, Gunma
  - Research Site, Ōta, Gunma
  - Research Site, Shibukawa, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Isehara, Kanagawa
  - Research Site, Sendai, Miyagi
  - Research Site, Sayama, Osaka
  - Research Site, Izumo, Shimane
  - Research Site, Mibu, Tochigi
  - Research Site, Shimotsuke, Tochigi
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Akita
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Ibaraki
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Nagasaki
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Murayama K, Kiguchi T, Izutsu K, Kameoka Y, Hidaka M, Kato H, Rai S, Kuroda J, Ishizawa K, Ichikawa S, Ando K, Ogura M, Fukushima K, Terui Y. Bendamustine plus rituximab in Japanese patients with relapsed or refractory diffuse large B-cell lymphoma. Ann Hematol. 2022 May;101(5):979-989. doi: 10.1007/s00277-022-04801-2. Epub 2022 Mar 4. PMID 35244756